CLINICAL TRIAL: NCT07374575
Title: Assessment of Knowledge, Attitudes, and Perceived Barriers Regarding the Oral Microbiome and Exosomes Among Egyptian Dental Professionals: A Cross-Sectional Questionnaire Study
Brief Title: Egyptian Dental Professionals' Perspectives on the Oral Microbiome and Exosomes
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adayil, Lecturer of Periodontology, Faculty of Dentistry, Cairo University , Cairo, Egypt, Cairo University
Other Study IDs: 10-2025
Record Dates: First submitted 2026-01-15; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Oral Health
Keywords: oral microbiome; exosomes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study employs a structured, validated questionnaire as the index test to objectively assess dental professionals' knowledge of the oral microbiome and exosomes, alongside attitudes, readiness, and perceived barriers. The primary aim is to develop and compare Microbiome Knowledge Scores (MKS) and Exosome Knowledge Scores (EKS) across dental specialties, workplace settings, and years of practice. Secondary aims include evaluating attitudes and perceived barriers, assessing the relationship between self-rated and objective knowledge, and identifying predictors of higher knowledge levels. The study tests the null hypotheses that MKS/EKS do not differ across demographic or practice characteristics and that self-rated knowledge does not correlate with objective knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Licensed dentists practicing in Egypt (general dentists and all specialties)
* age ≥18.

Exclusion Criteria:

* Undergraduate students/interns without a license
* dentists currently practicing abroad; duplicate entries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises licensed dentists practicing in Egypt, including general practitioners and all dental specialties, aged 18 years or older. Participants must hold a valid dental license and be actively practicing within Egypt. Excluded from the study are undergraduate dental students or interns without licensure, dentists currently practicing outside Egypt, and duplicate questionnaire responses.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Microbiome Knowledge Score (MKS) | 1 month
Exosome Knowledge Score (EKS) | 1 month